CLINICAL TRIAL: NCT01645111
Title: An Open-label Trial of Clevidipine for Controlled Hypotension During Spinal Fusion
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB12-00261
Record Dates: First submitted 2012-06-08; First posted 2012-07-20 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Neuromuscular Scoliosis
MeSH Terms: interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clevidipine (Active Comparator)
  Interventions: Drug: Clevidipine

INTERVENTIONS:
Drug: Clevidipine

SUMMARY:
The current study would prospectively evaluate the dosing requirements, efficacy and safety of clevidipine for controlled hypotension during spinal surgery in the pediatric population. As the investigators currently have projects underway which include those patients having scoliosis surgery for idiopathic scoliosis, this trial would include only those undergoing scoliosis surgery for neuromuscular disease.

DETAILED DESCRIPTION:
This would basically be an observational study without a significant change in our current practice. There would be no change in the standard and usual anesthetic care including premedication, anesthetic induction, intraoperative anesthetic management, and intraoperative monitoring. Our usual anesthetic routine includes:

1. Intravenous or oral premedication with midazolam
2. Inhalational or intravenous induction based on the preference of the patient
3. Facilitation of endotracheal intubation with a dose of rocuronium with placement of intraoperative monitors including an arterial cannula
4. Maintenance anesthesia to include desflurane titrated to maintain the bispectral index at 40-60, fentanyl 2-4 µg/kg followed by a remifentanil infusion to maintain the mean arterial pressure at 55-65 mmHg.
5. Tranexamic acid to limit intraoperative bleeding
6. As needed, agent to control blood pressure to maintain the MAP at 55-65 mmHg if remifentanil in doses up to 0.3 µg/kg/min are ineffective.

As needed, clevidipine will be started at 1 µg/kg/min and titrated up in 1 µg/kg/min every 1-2 minutes to achieve an MAP at 55-65mmHg. Vital signs including heart rate will be recorded every 1 minute until the target MAP is achieved and then at 15 minute increments after that.

ELIGIBILITY:
Inclusion Criteria:

* Spinal fusion for neuromuscular scoliosis.

Exclusion Criteria:

* Allergy to dihydropyridine calcium channel antagonists
* Allergy to soy or eggs
* Non-neuromuscular causes of scoliosis
* Disorders of lipid metabolism (clevidipine is in a lipid base)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Clevidipine: Clevidipine
Period: Overall Study
Arm/Group | Clevidipine
Started | 50
Completed | 35
Not Completed | 15
Not completed — Did not require Clevidipine | 15

BASELINE CHARACTERISTICS:
Arm/Group | Clevidipine
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 47
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve Target MAP
Description: The time between start of clevidipine infusion and patient reaching target mean arterial pressure (MAP) at 55-65 mmHg
Time Frame: First 30 minutes of infusion
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Clevidipine
Number analyzed (Participants) | 35
minutes | 9.2 (11.4)

ADVERSE EVENTS:
Arm/Group | Clevidipine
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes